CLINICAL TRIAL: NCT05161312
Title: Oncovox - An Acceptance and Commitment Therapy Guided Online Intervention to Improve Quality of Life in Breast Cancer Patients: a Randomised Clinical Trial
Brief Title: A Guided Online Intervention to Improve Quality of Life in Breast Cancer Patients - a Randomised Clinical Trial
Acronym: Oncovox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Silvia Nicolescu, Phd. Candidate, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BabesBolyaiOncovox
Record Dates: First submitted 2021-12-06; First posted 2021-12-17 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Cancer, Breast; Quality of Life; Distress, Emotional
Keywords: Acceptance and Commitment Therapy (ACT); Online intervention; Psychosocial intervention; Breast cancer; Quality of life; Randomized controlled trial
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iACT-BC: Oncovox experimental (Experimental): A guided internet-delivered ACT intervention to improve psychosocial outcomes in BCP diagnosed in the past two years.
  Interventions: Behavioral: iACT-BC: Oncovox
- Wait list control group (No Intervention): Wait list, treatment as usual

INTERVENTIONS:
Behavioral: iACT-BC: Oncovox — A guided internet-delivered ACT intervention to improve psychosocial outcomes in BCP diagnosed in the past two years
  Arms: iACT-BC: Oncovox experimental

SUMMARY:
Background: Online interventions can be a fast, cost-efficient, and convenient medium for providing breast cancer patients (BCP) with access to evidence-based interventions that address their emotional needs. As true as that may be, online interventions are still a novel research area that struggles in implementation.

Objectives: This study aims to determine the acceptability, feasibility, and efficacy of Oncovox, an iACT-BC, a guided internet delivered ACT intervention designed to improve psychosocial outcomes in BCP diagnosed within the last two years when compared to treatment as usual. The primary outcomes in this study are health related quality of life, behavioural activation, symptom interference and reward observation. The secondary outcomes are psychosocial distress, anxiety and depression and psychological flexibility.

Methods: A two-arm, parallel, open label, waiting list randomised controlled trial will investigate the effectiveness, feasibility, and acceptability of Oncovox.

Expected results: It is anticipated that Oncovox will show to be effective, feasible and acceptable programme in improving health related quality of life, behavioural activation, symptom interference, reward observation, psychological distress, anxiety, depression, and psychological flexibility in BCP diagnosed in the last two years, as opposing to a waiting list control under treatment as usual.

An exploratory moderator analysis will be employed to the assess the significance of Time x Group as well as Time x Group x Surgery type interactions for all outcome and process variables. A mediation analysis to assess the effect of psychological flexibility on the outcomes will also be applied.

The results of this research will be published in accordance with CONSORT 2010 and CONSORT-EHEALTH guidelines and should be available for publication in September 2022.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent.
* Age ≥ 18 years
* Ability to read and write in Romanian
* History of histologically or cytologically confirmed breast cancer
* An interval of < 24 months from histologically or cytologically confirmed breast cancer
* Ongoing curative cancer treatment
* Ongoing regular psychoactive medication only accepted if dosage has been stable during the last 3 months
* Daily access to the Internet by computer and/or smartphone
* Ability to use a computer and/or smartphone and the internet
* No participation on any other interventional study or clinical trial

Exclusion Criteria:

* Age ≤ 18 years
* Inability to co-operate and give informed consent
* Breast cancer not histologically or cytologically confirmed
* History of other malignancy within the last 5 years
* Current severe, uncontrolled systemic disease or mental disorder
* Absence of clinically significant symptoms
* Parallel ongoing psychological treatment
* Ongoing regular psychoactive medication if dosage has been changed during the last 3 months
* No access to the internet
* Inability to use a computer and/or smartphone and the internet
* Parallel ongoing participation in other interventional study or clinical trial
* Assessment by the investigator to be unable or unwilling to comply with the requirements of the protocol

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female BC diagnosis
Enrollment: 150 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Quality of life - Functional Assessment of Cancer Therapy - Breast (FACT-B) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  A a 37-item instrument designed to measure five domains of HRQOL in breast cancer patients: Physical, social, emotional, functional well-being as well as a breast-cancer subscale (BCS).
Behavioral activation - Behavioral activation scale (BAS) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  Assessing the appetitive-motivational system that is activated by reward consumption and conditioned signals of reward or non-punishment, triggering approach behaviour.
Symptom interference - MD Anderson Symptom Inventory (MDASI) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  Severity of symptoms experienced by patients with cancer and the interference with daily living caused by these symptoms.
Reward observation - Environmental reward observation scale (EROS) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  Reports on quantity and availability of reinforcement received by patient from environment

SECONDARY OUTCOMES:
Distress - Distress Thermometer (DT) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  a multifactorial unpleasant experience of a psychological (i.e., cognitive, behavioral, emotional), social, spiritual and/or physical nature that may interfere with the ability to cope effectively with cancer, its physical symptoms, and its treatment.
Anxiety & depression - Hospital Anxiety and Depression Scale (HADS) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  Measures anxiety and depression in a general medical population of patients
Psychological flexibility - Acceptance and Action Questionnaire for Cancer (AAQ-II-C) | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  Scale used to assess psychological inflexibility.

OTHER OUTCOMES:
Participants' attitudes towards internet interventions | Change from baseline to post-intervention (10 weeks after enrollment), Follow ups at 1, 2 and 12 months
  Attitudes towards internet interventions survey (ATTIS)
  Attitudes towards internet interventions survey (ATTIS)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia M Nicolescu, Ms, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No